CLINICAL TRIAL: NCT07380581
Title: The Herbal Acupoint Patch for Improving Pain, Depression, and Quality of Life in Dialysis Patient With Fistula-related Pain: Holistic Study for A Double-blind Randomized Controlled Trial
Brief Title: The Herbal Acupoint Patch for Dialysis Patient With Fistula-related Pain
Acronym: Fistula Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ming-Yen Tsai, Chief of Department of Chinese Medicine, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202302043A3C501; CORPG8N0441 (Other Grant/Funding Number: Chang Gung Memorial Hospital in Kaohsiung branch)
Record Dates: First submitted 2026-01-16; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: End Stage Chronic Renal Failure; Myofacial Pain
MeSH Terms: conditions — Renal Insufficiency, Chronic; Facial Pain | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham (No Treatment) (Sham Comparator)
  Interventions: Other: Sham (No Treatment)
- Artemisias-ginger patch (AGP) (Experimental)
  Interventions: Other: Artemisias-ginger patch (AGP)

INTERVENTIONS:
Other: Artemisias-ginger patch (AGP) — The TCM powder using extract powder that consists of Draconis Sanguis, Rz. Zingiberis Recens, and Artemisia princeps had been formulated into uniform 3X3 cm patch under the supervision of senior pharmacists. The 3 acupoints applied by study drug were LI 10, LU 5 and TE 5 with HD three times a week for 4 weeks.
  Arms: Artemisias-ginger patch (AGP)
Other: Sham (No Treatment) — The sham HAT was applied on 3 acupoints including LI 10, LU 5 and TE 5 with HD three times a week for 4 weeks.
  Arms: Sham (No Treatment)

SUMMARY:
To evaluate the effect of a traditional Chinese medicine (TCM) intervention on pain relief, mood and quality of life (QOL) in hemodialytic patients at a dialysis center in Southern Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* maintenance HD > 6 months ,
* reporting fistula pain during HD sessions that was associated with a hypersensitive palpable nodule in a taut band, at least 6 times in the past month,
* a NRS pain score >4,
* no changes in pain relievers such as NSAIDs, opioids, topical ointments, or muscle relaxants over the past week,
* voluntarily agreed to participate in the trial and presented written informed consent.

Exclusion Criteria:

* severe comorbid organ dysfunction,
* existence of cervical radiculopathy or thoracic outlet syndrome
* inflammation of the skin or soft tissue at the fistula site,
* dementia,
* psychiatric diseases,
* allergy to herbal patch
* currently participating in other clinical studies

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | Weeks 0 (baseline), 2, 4, and 6 (2 weeks of follow-up)
  Pain severity and interference are rated on a numerical rating scale (NRS) from 0 ("no pain"/"does not interfere") to 10 ("worst imaginable pain"/"completely interferes").

SECONDARY OUTCOMES:
Health Questionnaire Depression Rating Scale (PHQ-9) | Week 0 (baseline) and 4
  PHQ-9 is a 9-item, self-administered diagnostic tool used to screen for, diagnose, monitor, and measure the severity of depression in primary care and mental health settings. It scores symptoms based on the DSM-5 criteria over the past two weeks, with a total score ranging from 0 to 27.
EuroQol-5-dimension questionnaire (EQ-5D) | Week 0(baseline) and 4
  The EQ-5D consists of five dimensions that are rated on a 3-point scale, where lower scores indicate better health status

OTHER OUTCOMES:
Routine blood analysis | Week 0(baseline) and 4
  The outine blood analysis includes CBC, Kt/V, K, Ca, P, K, albumin, hsCRP, AST, and ALT.
Total number of analegics use in all HD sessions | Week 4
  Frequency of pain management including local analgesics, cryotherapy and oral painkillers during each dialysis was assessed within 12 sessions of study and was calculated by the number of participants in total.
Total number of early termination of hemodialysis | Week 4
  Total number of stopping the dialysis machine before the scheduled time (e.g., less than 4 hours) during 4-week treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital in Kaohsiung branch, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Data is being compiled and is expected to be submitted.